CLINICAL TRIAL: NCT07267832
Title: Impact of Health Promotion Service-Learning for Older Adults in Physiotherapy Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Collaborators: Hospital General Valencia (Other); Hospital Universitario La Fe (Other)
Responsible Party: Principal Investigator, Mercè Balasch i Bernat, Associate Professor, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: CEISH/47/2022
Record Dates: First submitted 2025-11-17; First posted 2025-12-05 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Healthy Students
Keywords: service-learning; physiotherapy; health promotion; teaching-learning methodology

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessor is blinded to participant group allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Service-Learning group (Experimental): Students work in groups to identify the needs of vulnerable older adults, researching and validating them with a mentor, combining individual and collaborative work, and culminating in the presentation and implementation of a health intervention, all accompanied by critical reflection on their personal and professional learning.
  Interventions: Other: health promotion through Service-Learning
- Traditional Learning group (Active Comparator): Students in the TL group follow a similar structure but do not engage directly with older adults. They identify needs solely through bibliographic research, review and discuss their findings with the teacher, and combine individual and group work. The intervention concludes with an oral presentation of the proposed health program to peers, illustrating it with examples.
  Interventions: Other: Health Promotion through Traditional Learning

INTERVENTIONS:
Other: health promotion through Service-Learning — Students of the Service-Learning Group (SLG) put their plans into practice by directly interacting with older adults in health centers, allowing them to observe needs firsthand and apply interventions in real-life contexts.
  Arms: Service-Learning group
Other: Health Promotion through Traditional Learning — Students in the Traditional Learning Group (TLG) develop their programs based solely on literature and research, without direct contact with patients. They analyze the needs of older adults through bibliographic sources, discuss their findings with the instructor, and integrate both individual and group work into their process. The TLG finalizes their project by presenting the proposed program to classmates, using examples to illustrate its application.
  Arms: Traditional Learning group

SUMMARY:
Currently, there is a lack of evidence regarding the impact of service-learning methodology (SL) on learning-related outcomes for physiotherapy students, specifically when designing and implementing health promotion programs for vulnerable older adults. The present study aims to compare the effects of an SL program versus a Traditional Learning (TL) approach on Basic Psychological Needs (BPN), motivation, academic engagement, and empathy in physiotherapy students.

This study is a randomized clinical trial. Eighty-three physiotherapy students are allocated to an SL group (SLG) or to a TL group (TLG). All students develop a health promotion and therapeutic exercise program for vulnerable older adults, in order to carry out prevention and health promotion activities. The SLG performs the program with real patients by visiting health centers, while the TLG does not meet real patients. BPN, motivation, academic engagement, and empathy, in their different dimensions, are evaluated pre- and post-intervention.

This study was registered retrospectively, as the recruitment and/or data collection had already started before registration.

DETAILED DESCRIPTION:
Health science professionals require both technical and interpersonal competencies to provide effective, patient-centered care. In physiotherapy, developing communication skills, empathy, and ethical awareness is essential for addressing patients' needs and situations of vulnerability. However, these interpersonal competencies are often insufficiently emphasized in traditional university curricula.

Service-Learning (SL) emerges as an innovative educational methodology that integrates academic learning with community service, allowing students to apply theoretical knowledge to real social contexts. Through direct engagement with community needs, SL promotes experiential learning, civic responsibility, and the development of transversal competencies such as empathy, communication, and teamwork. Aligned with the principles of the Self-Determination Theory, SL fosters the satisfaction of basic psychological needs-competence, autonomy, relatedness, and novelty-enhancing students' motivation and engagement.

Previous studies in health sciences suggest that SL improves academic performance, moral development, and self-determined motivation. In physiotherapy, it contributes to the acquisition of professional and interpersonal skills necessary for effective clinical practice. Nevertheless, there is limited evidence on the impact of SL when physiotherapy students design and implement health promotion programs for vulnerable older adults. Investigating this approach is therefore essential to understanding its potential to enhance learning outcomes and foster socially committed future professionals.

A randomized, assessor-blinded trial compares a Service-Learning (SL) intervention with a Traditional Learning (TL) approach in physiotherapy students. Eighty-three students from the University of Valencia (Spain) are randomly assigned to either the SL group (SLG, n=39) or the TL group (TLG, n=44).

The SL intervention follows six domains: (Domain 1) project introduction and formation of student groups; (Domain 2) identification of the physical, functional, and social needs of vulnerable older adults through direct contact and literature review; (Domain 3) discussion and validation of identified needs with mentor supervision; (Domain 4) autonomous individual work; (Domain 5) collaborative group work; and (Domain 6) final presentation in a clinical setting, including practical implementation with older adults and interactive discussion. Throughout all domains, students engage in guided critical reflection on the personal, professional, and social implications of their participation in the SL program.

The TL intervention consists of a parallel six-domain structure but without direct engagement with older adults: (Domain 1) project introduction and group formation; (Domain 2) identification of needs solely through bibliographic research; (Domain 3) review and discussion of findings with teacher supervision; (Domain 4) autonomous individual work; (Domain 5) collaborative group work; and (Domain 6) final oral presentation of the proposed health promotion program to peers at the university.

This study was registered retrospectively, as the recruitment and/or data collection had already started before registration.

ELIGIBILITY:
Inclusion Criteria:

* To be studying the Physiotherapy Degree in the Faculty of Physiotherapy of the University of Valencia.
* Willingness to participate

Exclusion Criteria:

* previous Service-Learning training

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2022-03-03 (Actual); Primary Completion 2022-04-17 (Actual); Study Completion 2022-04-17 (Actual)

PRIMARY OUTCOMES:
Basic Psychological Needs | baseline (pre-intervention) and immediately after the intervention
  The fulfillment of Basic Psychological Needs is measured using the Basic Psychological Need Satisfaction and Frustration Scale (BPNSNF), which evaluates the extent to which individuals experience satisfaction or frustration regarding four fundamental psychological needs: autonomy, competence, relatedness, and novelty. For each need, participants respond to items assessing both satisfaction and frustration on a 5-point Likert scale, where higher scores indicate greater satisfaction or greater frustration, respectively.

SECONDARY OUTCOMES:
Motivation | baseline (pre-intervention) and immediately after the intervention
  Motivation is assessed using the Scale of Motivation in Education, which includes 28 items across seven dimensions: Intrinsic Motivation - Knowledge, Intrinsic Motivation - Achievement, Intrinsic Motivation - Stimulating Experiences, Identified Regulation, Introjected Regulation, External Regulation, and Amotivation. Participants respond on a 7-point Likert scale, where 1 indicates "totally disagree" and 7 "totally agree." Higher scores in the first five dimensions indicate greater self-determined motivation, while higher scores in External Regulation and Amotivation reflect less self-determined forms of motivation.
Academic engagement | baseline (pre-intervention) and immediately after the intervention
  This outcome is measured using the short Spanish version of the Utrecht Work Engagement Scale, Student (UWES-S-9), an instrument described for analyzing engagement and widely used. This instrument measures three dimensions of academic engagement: vigor, dedication, and absorption. The scale consists of nine items in total, with three items corresponding to each dimension. Responses are rated on a 5-point Likert scale ranging from 1 (never) to 5 (always/every day). Higher scores indicate greater levels of academic engagement in each dimension.
Empathy | baseline (pre-intervention) and immediately after the intervention
  Empathy is evaluated using the Jefferson Scale of Physician Empathy (JSPE), a 20-item instrument scored on a 7-point Likert scale ranging from 1 (strongly disagree) to 7 (strongly agree). This scale is specifically designed to evaluate empathy within the context of patient care. It comprises three domains: (1) Empathic concern, which captures emotional sensitivity and concern for the patient's well-being; (2) Perspective taking, which reflects the ability to understand and consider the patient's viewpoint; and (3) Standing in the patient's shoes, which assesses the capacity to maintain appropriate emotional distance while still grasping the patient's experience. Higher scores across domains correspond to greater levels of empathy.

CONTACTS AND LOCATIONS:
Overall Officials: Mercè Balasch i Bernat, Principal Investigator — Department of Physiotherapy. Faculty of Physiotherapya. University of Valencia
Locations (1):
- Department of Physiotherapy. Faculty of Physiotherapy. University of Valencia, Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No